CLINICAL TRIAL: NCT00267943
Title: An Open-label Follow-up Trial of the Efficacy and Safety of Chronic Administration of the Fixed Dose Combination of Telmisartan 80 mg + Hydrochlorothiazide 25 mg Tablets Alone or in Combination With Other Antihypertensive Medications in Patients With Hypertension.
Brief Title: Open-label Follow-up Trial of Fixed Dose Combination of Telmisartan + Hydrochlorothiazide in Hypertensive Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 502.491
Record Dates: First submitted 2005-12-21; First posted 2005-12-22 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan; Hydrochlorothiazide

INTERVENTIONS:
Drug: telmisartan 80 mg + hydrochlorothiazide 25 mg

SUMMARY:
The primary objective is to assess the efficacy and safety of the fixed dose combination of telmisartan 80 mg + hydrochlorothiazide 25 mg (T80/H25) alone or in addition to other antihypertensive therapies during open-label, long-term treatment.

DETAILED DESCRIPTION:
Patients with a history of hypertension who completed a preceding trial (number 502.480) within the previous fourteen (14) days will be considered for entry to this long-term open-label trial. All patients will receive 'T80/H25'. Additional antihypertensive therapy will be allowed if the patients' blood pressure is not well controlled. [In the preceding double-blind trial 502.480, patients who failed to respond to the fixed dose combination of telmisartan 80 mg '+' hydrochlorothiazide 12.5 mg (T80/H12.5) were randomised to 'T80/H12.5' or T80H25 for eight weeks.] This is a multi-centre, multinational trial with approximately 80 study centres participating. Only study centres participating in the preceding trial 502.480 can enter patients into this open-label trial. It is anticipated that a maximum of 480 patients will be entered into the trial in seventeen countries. Each trial centre is expected to enter between four and twenty-four patients.

Enrollment of patients into this trial will finish when the last patient completes the preceding trial 502.480. At this time, centres will be notified of the termination of recruitment and will not be authorized to include any further patients.

Patients will visit the clinic one month, three months and six months later for assessment of their blood pressure and general health. Their participation in the study is complete six months after the start of the treatment period.

Study Hypothesis:

No statistical hypothesis will be tested. Descriptive statistics will be used to characterise the effects of treatment with T80/H25 with and without other antihypertensive treatments.

Comparison(s):

The proportion of patients achieving DBP control will be summarised by the total number of patients in the trial as well as by the maximum achieved dose level according to the two categories of T80/H25 alone (T80/H25) and with other antihypertensive medication added (T80/H25/other). An additional sub-group summary by the treatment group in the preceding trial 502.480 (T80/H12.5 and T80/H25) will also be presented.

ELIGIBILITY:
Inclusion criteria:

* Essential hypertension.
* Currently taking between one and three antihypertensive medications at a stable dose for at least four weeks before Visit 1 of preceding trial 502.480.
* Blood pressure not adequately controlled on existing treatment before entry to preceding trial 502.480 (inadequate control defined as seated DBP >= 95 mmHg on one current antihypertensive medication or DBP >= 90 mmHg on two or more current antihypertensive medications).
* Failure to respond to six weeks run-in treatment with T80/H12.5 in preceding trial 502.480. (Failure to respond defined as seated DBP >= 90 mmHg.)
* Willing and able to provide written informed consent.

Exclusion criteria:

* Women of child-bearing potential NOT practising acceptable means of birth control, positive serum pregnancy test, breastfeeding.
* Known or suspected secondary hypertension.
* Clinically significant change in ECG reported as adverse event in preceding trial 502.480.
* Any medical condition developing in preceding trial 502.480 that could be worsened by telmisartan/HCTZ (80/25).
* Discontinuation from preceding 502.480 trial for adverse event or any other reason.
* Mean SBP >= 200 mmHg.
* Severe hepatic or renal impairment.
* Bilateral renal artery stenosis (or in a solitary kidney), post-renal transplant or only one functioning kidney.
* Clinically relevant hypokalaemia or hyperkalaemia.
* Uncorrected volume or sodium depletion, primary aldosteronism.
* Hereditary fructose intolerance.
* Previous symptoms of angioedema after ACE inhibitors or angiotensin-II receptor antagonists.
* Drug or alcohol dependency within the six months prior to entry to 502.480. concurrent participation in another clinical trial or any investigational therapy.
* Hypertrophic obstructive cardiomyopathy, hemodynamically relevant stenosis of the aortic or mitral valve.
* Allergic hypersensitivity to any component of the formulations under investigation.
* Concomitant therapy with lithium, cholestyramine or colestipol resins.
* Non-compliance with study medication (less than 80% or more than 120%) during the preceding 502.480 trial.
* Any other clinical condition which, in the opinion of the investigator, would not allow safe administration of telmisartan or hydrochlorothiazide.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 639
Dates: Start 2006-01; Primary Completion 2007-01 (Actual); Study Completion 2007-01

PRIMARY OUTCOMES:
Proportion of patients achieving diastolic blood pressure (DBP) control 24 hours after last dose | at 6 months

SECONDARY OUTCOMES:
Change from baseline in trough seated DBP. | at 6 months
Change from baseline in trough seated systolic blood pressure (SBP) | at 6 months
Proportion of patients achieving DBP response (trough seated DBP<90 mmHg or trough seated DBP reduction from baseline ≥10 mmHg) | at 6 months
Proportion of patients achieving SBP response (trough seated SBP<140 mmHg or trough seated SBP reduction from baseline ≥10 mmHg) | at 6 months
Proportion of patients achieving SBP response (trough seated SBP<140 mmHg or trough seated SBP reduction from baseline ≥20 mmHg) | at 6 months
Proportion of patients in the trough seated BP category optimal | at 6 months
Proportion of patients in the trough seated BP category normal | at 6 months
Proportion of patients in the trough seated BP category high-normal | at 6 months
Proportion of patients in the trough seated BP category high | at 6 months
Proportion of patients requiring additional antihypertensive therapy to achieve DBP control | at 6 months
Additional reduction in BP by the use of additional antihypertensive therapy | at 6 months
Time to starting additional antihypertensive therapy | within 6 months
Incidence and intensity of Adverse events | 6 month
Physical examinations | 6 month
Change in laboratory parameters | 6 month
12-Lead Electrocardiogramm ECG | 6 month
Vital Signs (pulse rate, SBP, DBP) | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — BIL UK / Ireland
Locations (72):
- Denmark (5):
  - Boehringer Ingelheim Investigational Site, Birker?d
  - Boehringer Ingelheim Investigational Site, Haderslev
  - Boehringer Ingelheim Investigational Site, Odder
  - Boehringer Ingelheim Investigational Site, R?dovre
  - Boehringer Ingelheim Investigational Site, Vildbjerg
- Finland (3):
  - Boehringer Ingelheim Investigational Site, Helsinki
  - Boehringer Ingelheim Investigational Site, Joensuu
  - Boehringer Ingelheim Investigational Site, Turku
- France (3):
  - ALTI, Angers
  - Hopital Avicenne, Bobigny
  - Mg Recherches, Paris
- Germany (8):
  - Boehringer Ingelheim Investigational Site, Ellefeld
  - Boehringer Ingelheim Investigational Site, Flörsheim
  - Boehringer Ingelheim Investigational Site, Frankfurt am Main
  - Boehringer Ingelheim Investigational Site, Haag
  - Boehringer Ingelheim Investigational Site, Ingelheim
  - Boehringer Ingelheim Investigational Site, Nuremberg
  - Boehringer Ingelheim Investigational Site, Rodgau-Dudenhofen
  - Boehringer Ingelheim Investigational Site, Unterschneidheim
- Boehringer Ingelheim Investigational Site, Hong Kong, Hong Kong
- Ireland (7):
  - Boehringer Ingelheim Investigational Site, Birr
  - Boehringer Ingelheim Investigational Site, Carrigallen
  - Boehringer Ingelheim Investigational Site, Dublin
  - Boehringer Ingelheim Investigational Site, Gorey
  - Boehringer Ingelheim Investigational Site, Mallow
  - Boehringer Ingelheim Investigational Site, New Ross
  - Boehringer Ingelheim Investigational Site, Templeshannon
- Italy (4):
  - Ospedale Arnaboldi, Broni (pv)
  - Azienda Ospedaliera Universita di Ferrara, Ferrara
  - IRCCS San Raffaele, Roma
  - Ospedale Civile, Vittorio Veneto (tv)
- Boehringer Ingelheim Investigational Site, Kuching, Sarawak, Malaysia
- Netherlands (9):
  - Boehringer Ingelheim Investigational Site, Beerzeveld
  - Boehringer Ingelheim Investigational Site, Bennebroek
  - Boehringer Ingelheim Investigational Site, Ewijk
  - Boehringer Ingelheim Investigational Site, Hoogwoud
  - Boehringer Ingelheim Investigational Site, Nijverdal
  - Boehringer Ingelheim Investigational Site, Oude Pekela
  - Boehringer Ingelheim Investigational Site, Rijswijk
  - Boehringer Ingelheim Investigational Site, Roelofarendsveen
  - Boehringer Ingelheim Investigational Site, Rotterdam
- Norway (4):
  - Boehringer Ingelheim Investigational Site, Elverum
  - Boehringer Ingelheim Investigational Site, Moelv
  - Boehringer Ingelheim Investigational Site, Oslo
  - Boehringer Ingelheim Investigational Site, Skedsmokorset
- South Africa (8):
  - Boehringer Ingelheim Investigational Site, Bellville
  - Boehringer Ingelheim Investigational Site, Durban
  - Boehringer Ingelheim Investigational Site, Lenasia
  - Boehringer Ingelheim Investigational Site, Lenasia South
  - Boehringer Ingelheim Investigational Site, Midrand
  - Boehringer Ingelheim Investigational Site, Newtown
  - Boehringer Ingelheim Investigational Site, Pretoria
  - Boehringer Ingelheim Investigational Site, Soweto
- South Korea (2):
  - Boehringer Ingelheim Investigational Site, Incheon
  - Boehringer Ingelheim Investigational Site, Seoul
- Spain (8):
  - Hospital Municipal de Badalona, Badalona
  - Hospital de Galdakao, Galdakao / Vizcaya
  - Hospital Gral de Jerez de la Frontera, Jerez de La Frontera / Cadiz
  - C.A.P. Mosen Cinto Verdaguer, L'Hospitalet de Llobregat / Barcelona
  - Hospital Univ. Gregorio Mara?on, Madrid
  - C.A.P. Ronda Cerdanya, Mataro / Barcelona
  - Hospital de Mostoles - Medicina Interna, Mostoles / Madrid
  - Hospital del Conxo, Santiago de Compostela
- Sweden (4):
  - Boehringer Ingelheim Investigational Site, Eksjö
  - Boehringer Ingelheim Investigational Site, Karlstad
  - Boehringer Ingelheim Investigational Site, Uddevalla
  - Boehringer Ingelheim Investigational Site, Uppsala
- Switzerland (4):
  - Boehringer Ingelheim Investigational Site, Basel
  - Boehringer Ingelheim Investigational Site, Bellinzona
  - Boehringer Ingelheim Investigational Site, Saint-Imier
  - Boehringer Ingelheim Investigational Site, Vezia
- Boehringer Ingelheim Investigational Site, Taipei, Taiwan

REFERENCES:
- [Derived] Neldam S, Edwards C. Long-term, open-label evaluation of the safety and efficacy of telmisartan 80 mg/hydrochlorothiazide 25 mg fixed-dose combination alone or with other antihypertensive medication. Expert Opin Pharmacother. 2009 Feb;10(3):345-52. doi: 10.1517/14656560802707937. PMID 19191674